CLINICAL TRIAL: NCT02330913
Title: Novel Esophago-Jejunal Anastomosis Method During Totally Laparoscopic Total Gastrectomy: π-shape Esophagojejunostomy, Three-in-one Technique
Brief Title: Novel Esophago-Jejunal Anastomosis Method During Totally Laparoscopic Total Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Seung Wan Ryu, Director of Gastrointesinal surgery, associate professor, Keimyung University Dongsan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-11-001
Record Dates: First submitted 2014-12-19; First posted 2015-01-05 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Gastric Cancer
Keywords: total gastrectomy; intracorporeal; totally laparoscopic; esophagojejunostomy; anastomosis
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intracorporeal esophagojejunostomy (Experimental): Patient group with intracorporeal esophagojejunostomy with linear stapler
  Interventions: Procedure: Intracorporeal esophagojejunostomy

INTERVENTIONS:
Procedure: Intracorporeal esophagojejunostomy — Under laparoscopic view, esophagojejunostomy was pereformed with 60mm linear stapler on right side of distal esophagus like as functional end-to-end fashion before esophageal and jejunal resection. Then, three procedures of esophageal resection, common entry hole closure and jejunal resection was performed with a single use of 60mm stapler. Also, jejunojejunostomy was also performed via already made staple entry hole.

SUMMARY:
Laparoscopic gastrectomy became a good option for early gastric cancer. Surgical trend is gradually changed to totally laparoscopic gastrectomy from laparoscopy-assisted gastrectomy requiring mini-laparotomy. Various types of intracorporeal anastomosis have been introduced for esophagojejunostomy during total gastrectomy. We invented a novel anastomosis method using linear stapler for total gastrectomy. Three procedures (Jejunal resection, esophageal resection and closure of common entry hole after anastomosis) was performed with only one stapler. Therefore, the novel method is simple and fast. Also, this new technique is better economically than previously introduced anastomosis using linear stapler because lesser number of stapler is required. We want to demonstrate the feasibility of novel intracorporeal anastomosis method during laparoscopic total gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma in stomach
* Males or Females, aged≥20 years and ≤80 years
* Without serosa invasion, extraperigastric lymph node metastasis and other organ metastasis stage in preoperative evaluation, (cT1-3N0-1M0)
* Beyond the indication of ESD
* Tumor location in high body of stomach or requiring total gastrectomy
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1 at study entry
* American Society of Anesthesiolosists (ASA) score of 1 to 3
* The patient has given their written informed consent to participate in the study

Exclusion Criteria:

* Simultaneous malignancy in other organ
* Experience of previous laparotomy
* Experience of gastric resection including wedge resection
* Vulnerable subject

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-12; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Anastomosis related complication rate | During 30 days after operation
  Anastomotic leakage, intraluminal bleeding, or stenosis were considered as anastomosis related complication

CONTACTS AND LOCATIONS:
Overall Officials: Seung Wan Ryu, Ph.D., Principal Investigator — Keimyung University Dongsan Medical Center
Locations (1):
- Keimyung University Dongsan Medical Center, Daegu, South Korea